CLINICAL TRIAL: NCT03160690
Title: Changes in Choroidal Thickness After Non Penetrating Deep Sclerectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Pau Romera Romero (Unknown); Jorge Loscos Arenas (Unknown); Nevena Romanic Bubalo (Unknown); Jordi Castellví Manent (Unknown)
Responsible Party: Principal Investigator, Sandra Gómez Sánchez, Principal Investigator, Germans Trias i Pujol Hospital
Other Study IDs: OFT-ENP-2017-03
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Choroidal Thickness; Open Angle Glaucoma; Non Penetrating Deep Sclerectomy
Keywords: Choroidal thickness; Open Angle Glaucoma; Non penetrating deep sclerectomy
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Non penetrating deep sclerectomy — Non penetrating deep sclerectomy for open angle glaucoma

SUMMARY:
Prospective and observational study to determine if choroidal thickness increases after non penetrating deep sclerectomy in patients with open angle glaucoma

ELIGIBILITY:
Inclusion Criteria:

* Progressive Primary Open Angle Glaucoma

Exclusion Criteria:

* Age under 18yrs
* Myopia or Hyperopia higher than -6D or +6D
* Secondary glaucoma
* Ocular surgery other than cataract
* Other ocular pathology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with progressive open angle glaucoma although topical treatment with indication for non penetrating deep sclerectomy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-06-17 (Estimated); Primary Completion 2017-11-17 (Estimated); Study Completion 2018-05-17 (Estimated)

PRIMARY OUTCOMES:
Change in Choroidal thickness | before and 1 week, 1 month, 3 months and 6 months after non penetrating deep sclerectomy
  Choroidal thickness measured by optic coherence tomography
Change in Intraocular pressure | before and 1 week, 1 month, 3 months and 6 months after non penetrating deep sclerectomy
  mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Gómez Sánchez, MD, Principal Investigator — Germans Trias i Pujol Hospital; Pau Romera Romero, MD, Principal Investigator — Germans Trias i Pujol Hospital; Jorge Loscos Arenas, PhD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No